CLINICAL TRIAL: NCT06719193
Title: Demonstrating Multipronged and Optimized Novel Strategies to Reinforce Actions Targeted At Eliminating Tuberculosis (DeMONSTRATE-TB): a Sequential Exploratory Mixed Method Study in Ethiopia
Brief Title: DeMONSTRATE-TB Study in Ethiopia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Management Sciences for Health (Other)
Collaborators: KNCV Tuberculosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 37.2022; 72066320CA00009 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Reducing Tuberculosis Incidence
Keywords: tuberculosis prevalence; tuberculosis incidence; tuberculosis elimination; tuberculosis preventive therapy; quasi experimental; ethiopia

STUDY DESIGN:
Intervention Model Description: A sequential exploratory mixed-method study with a dominant controlled before-after (or quasi-experimental) design will be the main design of this study, followed by qualitative methods. The aim of the qualitative component is to explore whether the ETB intervention package is feasible and helps achieve TB elimination in Ethiopia. In-depth interviews (IDIs) and focus-group discussions (FGDs) with TB program managers and health extensions workers, community leaders, and selected heads of households involved the study will be conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced community-wide TB intervention (Experimental): Enhanced community-wide TB intervention strategy with intensive screening and health education
  Interventions: Combination Product: Enhanced community-wide TB intervention
- Routine TB program activities (Active Comparator): TB standard of care per Ethiopia's national guidelines
  Interventions: Combination Product: Routine TB program activities

INTERVENTIONS:
Combination Product: Enhanced community-wide TB intervention — Interventions in the intervention arms consist of the following key components:
  1. an optimized national recommended set of interventions; such as the implementation of all types of contact investigation, targeted TB screening and diagnosis at key affected population, and optimized HIV screening and TPT for PLHIV;
  2. intensive, active, and community-based HH screening and diagnosis of TB using combined TB screening (clinical and X-ray) and X-pert MTB/RIF, as indicated;
  3. community-based enhanced TPT; and
  4. community-based awareness creation and health education using the community social associations.
  Arms: Enhanced community-wide TB intervention
Combination Product: Routine TB program activities — In the control arm, the standard of care will continue per the national guideline.
  Arms: Routine TB program activities

SUMMARY:
Ending the TB epidemic by 2035 in Ethiopia would be possible if TB notification declines by an annual factor of at least 15% from the current notification rate of 132 per 100,000 population. This requires highly effective strategies to reduce TB transmission and maximize TB prevention among populations at risk of developing TB, such as Household contacts and people living with HIV.

The investigators hypothesize that community wide administration of enhanced TPT will accelerate decline in TB incidence rates when combined with an optimized currently recommended comprehensive TB prevention and care packages described below. The investigators further hypothesize that such intervention packages will be acceptable to the community, providers and policy makers, and that they will be cost-effective.

Based on the study results, a TB elimination framework in high burden TB regions and woredas in Ethiopia will be developed, and local evidence to enhance the shift toward TB elimination will be provided as input to the appropriate allocation of resources.

ELIGIBILITY:
Inclusion Criteria:

1. Adults:

   * Greater than or equal to 18 years old
   * Provides consent
   * Living in study site area (woreda)
2. Children

   * Aged 12 to 17 years
   * Living in the study site area (woreda)
   * Assent to enrollment
   * Guardian provides consent for enrollment
3. Younger children:

   * Less than 12 years old
   * Living in the study site area (woreda)
   * Consent for enrollment provided by the guardian

Exclusion Criteria:

1. Adults:

   * Does not provide consent
   * Declines to provide contact information
   * Less than 18 years
   * Living outside of the study site area
   * Declines to allow study staff to contact them by phone and in person if they miss a study visit
2. Children

   * Does not provide assent
   * Guardian does not provide consent
   * Guardian declines to provide contact information
   * Not within 12 to 17 years
   * Living outside of the study site area
   * Guardian declines to allow study staff to contact them by phone and in person if they miss a study visit
3. Younger Children

   * Guardian does not provide consent
   * Guardian declines to provide contact information
   * Not less than 12 years
   * Living outside of the study site area
   * Guardian declines to allow study staff to contact them by phone and in person if they miss a study visit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 131438 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Population-level TB prevalence | Semi-annual screening (up to 2 years)
  Demonstrate the impact and feasibility of a community wide TPT in reducing TB incidence when administered in combination with intensified active TB case finding, improved diagnostic capacity, and general awareness creation. Ultimately, the evidence generated will be used to develop a TB elimination framework for broader application.

SECONDARY OUTCOMES:
Change in TB treatment outcomes | Baseline and at 2 years
  TB treatment outcomes are classified as cured, treatment completed, treatment failure, died, loss-to-follow up, and not evaluated based on the World Health Organization (WHO) definition and reporting framework for tuberculosis. Baseline TB treatment outcome will be collected at the start through a baseline prevalence survey to understand the baseline status of TB outcomes. This data on TB treatment outcomes will then be compared after two years of intervention in both intervention and control woredas to understand if there is an improvement in favorable TB treatment outcomes (i.e., cured or treatment completed) and decrease in less favorable TB treatment outcomes (i.e., treatment failed, died, loss-to-follow up) in the intervention sites compared to the standard of care control sites.

OTHER OUTCOMES:
Improved Knowledge, attitude and practices (KAP) regarding tuberculosis among participants in intervention sites (woredas). | Baseline and at 2 years
  The tuberculosis (TB) knowledge, attitude and practices (KAP) survey tool (both open and close ended questions) will be administered at baseline and at year two to measure health seeking behaviors, TB knowledge and awareness, TB attitudes and care-seeking behaviors, TB attitudes and stigma, and TB awareness and sources of information among the participants in the intervention sites and control sites. The investigators will compare improvements in reports of knowledge from the KAP survey tool between baseline and at 2 years across both the control and intervention sites to understand if there are higher improvements at the intervention sites.

CONTACTS AND LOCATIONS:
Locations (2):
- Ethiopia (2):
  - Gedebe Hassassa woreda, West Arsi Zone, Ormoia Regional State
  - Boloso Bombe woreda, Wolayita Zone, South Ethiopia Regional State

IPD SHARING:
Plan to Share IPD: No